CLINICAL TRIAL: NCT04562857
Title: Effects of Exercise Training in Patients With Atrial Fibrillation and Sleep Apnea: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Swinburne University of Technology (Other); National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physical therapy for cardiopulmonary disorders, Faculty of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF and sleep apnea
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obstructive sleep apnea (Active Comparator): interval exercises (intervention) on bicycle for patients with AF and OSA for 10 weeks, 3 times/week for duration of 30-45 min/ session.
  Interventions: Behavioral: Moderate intensity interval training (MITT)
- Central sleep apnea (Active Comparator): interval exercises (intervention) on bicycle for patients with AF and CSA for 10 weeks, 3 times/week for duration of 30-45 min/ session.
  Interventions: Behavioral: Moderate intensity interval training (MITT)

INTERVENTIONS:
Behavioral: Moderate intensity interval training (MITT) — interval exercises (intervention) on bicycle for patients with AF and OSA or AF with CSA for 10 weeks, 3 times/week for duration of 30-45 min/ session.

SUMMARY:
Background: There are still many gaps in research concerning the effect of different physical training modalities on sleep deprivation in the population with different types of sleep apnea. Aims: The purpose of this study was to examine the effect of moderate-intensity interval training (MITT) on patients with different types of sleep apnea.

DETAILED DESCRIPTION:
Methods: 15 Participants aged 45-65 years were randomized into two groups: obstructive sleep apnea group (OSA), and central sleep apnea group (CSA). The training lasted ten consecutive weeks with 30 uninterrupted sessions. The actigraph together with the Pittsburg sleep quality index (PSQI) was used in sleep quality assessment. The actigraph (Actiwatch Minimitter Company, Incorporated (INC) - Sunriver, OR, USA) was placed on the non-dominant wrist and activities were monitored continuously while being recorded at one-minute intervals. The participants kept the device for a period of 96 hours, filled PSQI, and did 6MWT before the first and last training sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have AF confirmed by ECG
2. Their ages range from 45 and 65 years of age
3. Medically stable patients.
4. Current complaint of poor Sleep quality (SQ) (score > 5 of the SQ scale)
5. Patients who have OSA or CSA confirmed by polysomnography

Exclusion Criteria:

* Any patient was known to have any unstable medical condition;or with any known musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise, was excluded from the study.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Sleep quality scores (0 is best, 3 is worst) | 10 weeks
  data about sleep from Pittsburgh sleep quality index questionnaire
sleep latency (in min) | 10 weeks
  time spent in bed before falling asleep (from the actigraph)
Total sleep time (in hours) | 10 weeks
  Total time actually slept (from the actigraph)
Sleep fragmentation index (in %) (the more means worse) | 10 weeks
  Index of the level of the sleep continuity (from the actigraph)
cutpoints | 10 weeks
  numbers displayed on the actigraph to give a picture about activity level

SECONDARY OUTCOMES:
six minute walking distance (in meters) | 10 weeks
  represent aerobic capacity (distance walked in 6 min)

CONTACTS AND LOCATIONS:
Overall Officials: Hady Balabel, Principal Investigator — Cairo University
Locations (1):
- National heart institute, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for12 months
Access Criteria: will upload it to the journal of publication

DOCUMENTS (1):
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT04562857/ICF_000.pdf